CLINICAL TRIAL: NCT01106235
Title: Phase I Study To Evaluate Cellular Adoptive Immunotherapy Using Autologous IL-21 Modulated CD8+ Antigen-Specific T Cells For Patients With Metastatic Melanoma
Brief Title: Therapeutic Autologous Lymphocytes, Cyclophosphamide, and Aldesleukin in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Yee, Cassian, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2390.00; NCI-2010-00146 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-04-08; First posted 2010-04-19 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (immunostimulant, autologous lymphocytes, and chemo) (Experimental): Patients receive cyclophosphamide IV on days -3 and -2 followed by an infusion of IL-21 modulated, MART-1 specific CD8+ cytotoxic T lymphocytes over 30-60 minutes on day 0. Beginning within 24 hours of T cell infusion, patients receive low-dose aldesleukin SC BID for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: therapeutic autologous lymphocytes; Biological: aldesleukin; Drug: cyclophosphamide; Procedure: biopsy

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Given IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies

SUMMARY:
RATIONALE: Aldesleukin may stimulate lymphocytes to kill melanoma cells. Treating lymphocytes with interleukin-21 in the laboratory may help the lymphocytes kill more tumor cells when they are put back in the body. Giving therapeutic autologous lymphocytes together with cyclophosphamide and aldesleukin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of giving therapeutic autologous lymphocytes together with cyclophosphamide and aldesleukin in treating patients with metastatic melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and toxicity of adoptively transferred interleukin (IL)-21 modulated cytotoxic T-lymphocyte (CTL) targeting a melanoma associated antigen in patients following cyclophosphamide conditioning.

II. Evaluate the functional and numeric in vivo persistence of adoptively transferred IL-21 modulated CTL and factors contributing to immunopotentiation in patients receiving IL-21 modulated CTL following cyclophosphamide conditioning.

SECONDARY OBJECTIVES:

I. Evaluate the antitumor effect of adoptively transferred IL-21 modulated CD8+ antigen-specific CTL following cyclophosphamide conditioning and post-infusion IL-2.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) on days -3 and -2 followed by an infusion of IL-21 modulated, melanoma antigen recognized by T cell (MART)-1 specific CD8+ cytotoxic T lymphocytes over 30-60 minutes on day 0. Beginning within 24 hours of T-cell infusion, patients receive low-dose aldesleukin subcutaneously (SC) twice daily (BID) for 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 8-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* FOR LEUKAPHERESIS:
* Pulse > 45 or < 120
* Weight >= 45 kg
* Temperature =< 38 Celsius (C) (=< 100.4 Fahrenheit [F])
* White blood cells (WBC) >= 3000
* Hematocrit (HCT) >= 30%
* Platelets >= 100,000
* FOR T CELL INFUSION:
* Histopathological documentation of melanoma concurrent with the diagnosis of metastatic disease
* Tumor expression of MART-1 (2+ staining or > 25%) by immunohistochemistry (IHC)
* Able to tolerate high-dose cyclophosphamide
* Expression of human leukocyte antigen (HLA)-A2
* Zubrod performance status of 0-1
* Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray, computed tomography [CT] scan)
* Normal cardiac stress test within 182 days prior to enrollment is required of all patients over 50 years old or those with an abnormal electrocardiogram (ECG), any history of cardiac disease, a family history of cardiac disease or hypertension

Exclusion Criteria:

* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to entry
* Serum creatinine > 1.6 mg/dL or creatinine clearance (CrCl) < 75 ml/min (calculated: Cockcroft and Gault equation: CrCl = (140 - age) x ideal body weight (IBW)/(serum creatinine [Scr] x 72) (x 0.85 for females)
* Serum glutamic oxaloacetic transaminase (SGOT) > 150 IU or > 3 x upper limit of normal
* Direct bilirubin > 1.0 mg/dL
* Prothrombin time > 1.5 x control (in the absence of systemic anticoagulation)
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing at the discretion of their primary physician
* Significant cardiovascular abnormalities as defined by any one of the following:
* Congestive heart failure,
* Clinically significant hypotension,
* Symptoms of coronary artery disease,
* Presence of cardiac arrhythmias on electrocardiogram (EKG) requiring drug therapy
* Symptomatic central nervous system metastases greater than 1 cm at time of therapy; patients with 1-2 asymptomatic, less than 1cm brain/central nervous system (CNS) metastases without significant edema may be considered for treatment; if sub-centimeter CNS lesions are noted at study entry, then a repeat imaging will be performed if more than 3 weeks have elapsed from the last scan; patients will not be treated if CNS lesions are > 1 cm or if patient is symptomatic from brain metastasis
* Patients with active infections or oral temperature > 38.2 C within 72 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy
* Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 3 weeks prior to T cell therapy; (patients with bulky disease may undergo cytoreductive chemotherapy but treatment will be discontinued at least 3 weeks prior to T cell therapy)
* Clinically significant autoimmune disorders or conditions of immunosuppression; patients with acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV)-1 associated complex or known to HIV antibody seropositive or known to be recently polymerase chain reaction positive (PCR+) for hepatitis are not eligible for this study; virology testing will be done within 6 months of T cell infusion; the severely depressed immune system found in these infected patients and the possibility of premature death would compromise study objectives
* Patients who, in the opinion of their physician, are not clinically suited for high-dose cytoxan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 | 10 weeks post infusion
Functional and numeric in vivo persistence of adoptively transferred IL-21 modulated CTL and factors contributing to immunopotentiation in patients receiving IL-21 modulated CTL following cyclophosphamide conditioning | 10 weeks post infusion
  Descriptive statistics (average, median standard deviation and student's t test) will be used to determine if an increase in the duration of in vivo persistence is observed using IL-21 modulated T cells when retrospectively compared with T cells generated under standard culture conditions (no IL-21 exposure in vitro).

SECONDARY OUTCOMES:
In vivo persistence and anti-tumor effect of the infused IL-21 modulated CTL | 10 weeks post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States